CLINICAL TRIAL: NCT04183101
Title: Phase 2, Multicenter, Randomized, Open-label, Controlled, 2-arm Cross-over Study to Evaluate the Clinical Efficacy of a Renin Inhibitor, Aliskiren, Compared to an Angiotensin Converting Enzyme Inhibitor, Enalapril, in C3 Glomerulopathy
Brief Title: Evaluation of a Renin Inhibitor, Aliskiren, Compared to Enalapril, in C3 Glomerulopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001440-22; 2019-001440-22 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-12-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: C3 Glomerulopathy; Membranoproliferative Glomerulonephritis; Complement Abnormality; Dense Deposit Disease; C3 Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — aliskiren; Enalapril

STUDY DESIGN:
Intervention Model Description: Phase 2, multicenter, randomized, open-label, controlled, 2-arm cross-over study to evaluate the clinical efficacy and safety of a renin inhibitor, aliskiren, compared to an angiotensin converting enzyme inhibitor, enalapril, in children and adults with C3 glomerulopathy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aliskiren treatment (Experimental): Patients will be randomized to tablet treatment with aliskiren (target daily dose) 150-300 mg once daily or every other day (depending on weight) for 6 months. After 6 months the patients will be switched to tablet treatment with enalapril (target daily dose 7.5-20 mg once or twice a day) for the coming 2,5 years.
  Interventions: Drug: Aliskiren
- Enalapril treatment (Active Comparator): Patients will be randomized to tablet treatment with enalapril (target daily dose 7.5-20 mg once or twice a day) for 6 months. After 6 months the patients will be switched to tablet treatment with aliskiren (target daily dose) 150-300 mg once daily or every other day (depending on weight) for the coming 2,5 years.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Aliskiren — Patients will be randomized to start treatment with aliskiren tablet 150 mg every other day up to 300 mg daily depending on weight. After 6 months switch to enalapril 2.5-20 mg daily and continue with that 2.5 years.
  Other Names: Enalapril
  Arms: Aliskiren treatment
Drug: Enalapril — Patients will be randomized to start with enalapril 2.5-20 mg daily depending on weight. After 6 months switch to aliskiren tablet 150 mg every other day up to 300 mg daily depending on weight and continue with this treatment for 2.5 years.
  Other Names: Aliskiren
  Arms: Enalapril treatment

SUMMARY:
The aim of this cross-over trial is to assess aliskiren, a direct renin inhibitor, as a novel treatment to block complement activation in the kidneys and thereby attenuate renal disease and stabilize or improve kidney function and compare it to the currently used treatment with the angiotensin converting enzyme inhibitor, enalapril, in patients with the complement-mediated renal disease C3 glomerulopathy. Patients will be randomized to one or the other treatment for the first 6 months and then switch to the other treament for the following 2.5 years. Treatment will continue for altogether 3 years for each patient.

DETAILED DESCRIPTION:
The primary objective is to assess the effect and safety of aliskiren on reducing systemic and local complement activation as indicated by a reduction of serum C3 during the cross-over study and serum C3 and complement deposition in renal biopsies during the extension study in patients with C3 glomerulopathy as compared to the currently used treatment with the angiotensin converting enzyme inhibitor (ACEi) enalapril.

Secondary objectives are to assess the effect of aliskiren as compared to the currently used treatment with the ACEi enalapril on: complement activation (such as serum C3a, C3dg, C5a and related complement assays), proteinuria, kidney function, kidney biopsy findings, blood pressure, activation of the renin angiotensin system.

Aliskiren will be administered orally in tablet form at 150 -300 mg/daily (maximal dose 300 mg). Enalapril 2.5-20 mg/daily (maximal dose 20 mg). These drugs may be administered once or twice.

The investigators estimate an inclusion of maximum 15 patients for start of treatment with aliskiren and maximum 15 patients for start of treatment with enalapril. Suitable patients will be chosen from those patients who:

1. Do not have severe renal failure. Pediatric patients will be included if they have a glomerular filtration rate ≥ 50 ml/min/1.73m2, adults ≥ 30 ml/min/1.73m2.
2. Children, above the age of 6 years of age and adults.
3. Patients treated with aliskiren will be compared to patients treated with the ACE inhibitor enalapril as monotherapy. Use of ACE inhibitor as a nephroprotective therapy will increase renin levels without blocking its effect. Thus, the investigators will compare patients on aliskiren with those on enalapril to investigate if ACE inhibition as monotherapy has a negative effect on complement activation in comparison to direct renin inhibition.
4. Patients treated with immune suppressive medications at the start (such as mycophenolate mofetil (MMF) or corticosteroids) will be compared to patients treated with MMF or steroids plus aliskiren or enalapril.

All suitable patients who fulfill inclusion criteria and who submitted written informed consent (patient or patient's legal guardians) will have undergone a renal biopsy at the most 2 years before inclusion or at inclusion and will be randomized for treatment with aliskiren or enalapril. After 6 months patients on aliskiren will switch to enalapril and vice versa, patients on enalapril will switch to aliskiren treatment. Patients will be followed routinely, every 3rd month, regarding renal function (creatinine, urea, estimated glomerular filtration rate), albumin (blood and urine), renin levels and complement activation assays in blood samples (C3, C3dg, C5, properdin, soluble terminal complement complex, C3a, C5a, C3 nephritic factor and other complement assays). The follow-up period, a total of 3 years from the start, will be carried out by the patient's own nephrologist and will not differ from the clinical follow-up offered patients not participating in the study. After 1-3 years (when medically indicated but at the most 3 years after start), a repeat renal biopsy will be performed to validate the effect of treatment on renal morphology. Renal biopsies, both the initial and the repeat biopsy, will be evaluated for complement deposition and glomerular basement membrane thickness.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≥ 6 years and adults.
2. Initial diagnosis of Dense Deposit Disease and C3 glomerulonephritis confirmed by kidney biopsy obtained not more than 2 years before the first dose of the study drug.
3. Either absence of treatment at the study start or ongoing treatment with aliskiren, angiotensin converting enzyme inhibitors, angiotensin receptor blockers or immune suppressive medications (such as mycophenolate mofetil/MMF or corticosteroids)
4. Written informed consent has been given by:

   1. the patient's legal guardians if the patient is less than 15 years old
   2. the patient and his/her legal guardians if the patient is ≥ 15 but < 18 years old
   3. the patient, if the patient is ≥ 18 years old
5. Female subjects of childbearing potential must:

   1. Understand that the study medication is expected to have a teratogenic risk
   2. Agree to use a highly effective contraceptive during study drug therapy. This applies unless the subject is less than 18 years of age, has not had sexual debut and commits to sexual abstinence confirmed by a pregnancy test on every study visit. Either of the following methods of contraception may be used:

      * Combined (estrogen and progesterone) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal
      * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable or implantable
      * Intrauterine device
      * Intrauterine hormone-releasing system
      * Bilateral tubal occlusion
      * Vasectomized partner
      * Sexual abstinence
      * Male or female condom with or without spermicide
      * Cap, diaphragm or sponge with spermicide
   3. Agree to have a pregnancy test before the start of study medication. This requirement also applies to women of childbearing age who practice complete and continued abstinence and adolescent girls after menarche.
   4. Agree to have a pregnancy test every 3rd month including at the end of study treatment, except in the case of confirmed tubal sterilization. This requirement also applies to women of childbearing age who practice complete and continued abstinence and adolescent girls after menarche.

Exclusion Criteria:

1. Known allergy to aliskiren, ACEi or substances contained in these preparations.
2. Angioedema caused by aliskiren or enalapril
3. Weight < 25 kg
4. Glomerular filtration rate ≤ 50 ml/min/1.73 m2 (measured by iohexol clearance) in children and ≤ 30 ml/min/1.73 m2 in adults.
5. Rapid deterioration of kidney function during the latest year of the disease
6. Patients with a renal transplant
7. Immune complex-mediated membranoproliferative glomerulonephritis (such as in HIV infection, hepatitis, SLE)
8. Females who breastfeed, are pregnant or planning to become pregnant during the study.
9. Co-morbidity such as malignancy, congestive heart failure, recent myocardial infarction.
10. Mental incapacity or language barriers to understand the contents of the study design.
11. Simultaneous use of another complement-antagonist (such as eculizumab). Eculizumab must be discontinued and complement activity normalized before the start of study drug.
12. Simultaneous use of aliskiren or enalapril with cyclosporine or nonsteroidal anti-inflammatory drugs (NSAID).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
C3 levels in serum | 3 years
  To assess the effect and safety of aliskiren as compared to enalapril on reducing systemic complement activation as assayed by C3 levels in serum.
Complement deposition in kidneys | 3 years
  To quantify complement deposition in kidney biopsies from patients with C3 glomerulopathy using immunohistological staining

SECONDARY OUTCOMES:
C3a in serum | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on C3a in serum
C3dg in plasma | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on C3dg in plasma
C5a in serum | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on C5a in serum
Glomerular basement membrane thickness | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on glomerular basement membrane thickness assessed by electron microscopy measurement
Proteinuria | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on protein levels in urine measured as the ratio between albumin/creatinine in urine

OTHER OUTCOMES:
Renal function | 3 years
  To assess the effect of aliskiren compared to currently used treatment with the ACEi enalapril on kidney function measured as iohexol clearance glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Diana Karpman, Principal Investigator — Region Skåne
Locations (4):
- Sweden (4):
  - Sahlgrenska Hospital, Gothenburg
  - Region Skåne Skåne Universitetssjukhus, Lund
  - Karolinska Hospital, Stockholm
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
The study and de-identified data will be shared with study coordinators at various sites
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years from the start, two years of inclusion until the inclusion of the last patient
Access Criteria: Data will be presented at meetings and by de-identified emails

REFERENCES:
- [Background] Bekassy ZD, Kristoffersson AC, Rebetz J, Tati R, Olin AI, Karpman D. Aliskiren inhibits renin-mediated complement activation. Kidney Int. 2018 Oct;94(4):689-700. doi: 10.1016/j.kint.2018.04.004. Epub 2018 Jun 5. PMID 29884545
- [Background] Smith RJH, Appel GB, Blom AM, Cook HT, D'Agati VD, Fakhouri F, Fremeaux-Bacchi V, Jozsi M, Kavanagh D, Lambris JD, Noris M, Pickering MC, Remuzzi G, de Cordoba SR, Sethi S, Van der Vlag J, Zipfel PF, Nester CM. C3 glomerulopathy - understanding a rare complement-driven renal disease. Nat Rev Nephrol. 2019 Mar;15(3):129-143. doi: 10.1038/s41581-018-0107-2. PMID 30692664
- [Background] Taal MW, Brenner BM. Renoprotective benefits of RAS inhibition: from ACEI to angiotensin II antagonists. Kidney Int. 2000 May;57(5):1803-17. doi: 10.1046/j.1523-1755.2000.00031.x. PMID 10792600